CLINICAL TRIAL: NCT06331247
Title: MIND Diet to Improve Cognitive Function in Mild Stroke Patients (MINDICOMS) II: A Pilot Randomized Control Trial
Brief Title: MIND Diet to Improve Cognitive Function in Mild Stroke Patients (MINDICOMS) II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Changzheng Yuan, Research Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20230520-2
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Stroke; Cognitive Change; Cerebrovascular; Disorder, Thrombotic
Keywords: Stroke; Cognitive Change; MIND diet; Dietary pattern
MeSH Terms: conditions — Dementia; Stroke

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel design, with one arm being the control arm (usual medical care) and the other being the intervention arm (MIND diet intervention + usual medical care).
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be masked from the assignment of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): Usual medical care (including general dietary advice).
  Interventions: Behavioral: General dietary advice; Other: Routine medical care
- MIND diet intervention arm (Active Comparator): Usual medical care (including general dietary advice) plus the MIND diet intervention.
  Interventions: Behavioral: General dietary advice; Behavioral: Localized MIND diet intervention; Other: Routine medical care

INTERVENTIONS:
Behavioral: General dietary advice — General dietary advice according to the Chinese Dietary Guidelines 2022.
Behavioral: Localized MIND diet intervention — The MIND diet intervention, composed of the consumption of whole grains, dark green leafy vegetables, dark red/yellow vegetables, other vegetables, berries and citrus, poultry, fish and seafoods, beans and legume, nuts, olive and seed oils, and green tea, and restricting red and processed meats, animal fat, fried foods, and sweets and pastries.
  Arms: MIND diet intervention arm
Other: Routine medical care — Routine medical care and follow-ups.

SUMMARY:
A 6-month pilot randomized controlled trial designed to test the effect of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet + usual medical care versus usual medical care on cognitive change and several other secondary outcomes through a randomized controlled trial in 60 mild stroke patients aged 35-70 years without dementia.

DETAILED DESCRIPTION:
Mediterranean-DASH (Dietary Approach to Stop Hypertension) Intervention for Neurodegenerative Delay (MIND) Diet and Cognitive Decline in Mild Stroke Patients (MINDICOMS) II is a 6-month pilot randomized controlled trial designed to test the effects of the MIND diet on cognitive change and several other secondary outcomes among 60 individuals aged 35-70 years without dementia. The proposed MIND diet for this study is a hybrid of the Mediterranean and DASH diets but with selected modifications based on the most compelling evidence in the diet-dementia field and Chinese Dietary Guidelines 2022. Specifically, the proposed MIND diet will emphasize the consumption of whole grains, dark green leafy vegetables, dark red/yellow vegetables, other vegetables, berries and citrus, poultry, fish and seafood, beans and legume, nuts, olive and seed oils, and green tea, and restrict red and processed meats, animal fat, fried foods, and sweets and pastries. The trial will employ a parallel group design comparing the effects on global cognitive change of the MIND intervention diet to usual medical care among 60 mild stroke patients aged 35-70 years. Secondary outcomes will include cognitive function changes in several domains, brain imaging marker changes, dietary behaviour changes, daily living behaviour ability changes, mental health changes, and plasma biomarker changes. In addition, this trial will examine potential effect mediators and modifiers. The proposed study is sited at the Bo'Ao District, Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou. Specialized laboratories will conduct biochemical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed new cerebral infarction, onset hospitalization time ≤14 days
* National Institutes of Health Stroke Scale (NIHSS) score of 0-6, with no difficulty in autonomous eating or aphasia
* Baseline MMSE score being 16-25/30 points or MoCA score ≤24/30 points, with signs of post-stroke cognitive decline
* Baseline MIND dietary pattern screening scale score ≤10/15 points
* Body mass index no less than 18.0 kg/m2
* Normal chewing function, able to eat hard foods such as nuts
* Willing to participate and sign an informed consent form
* Agree not to take over-the-counter nutritional supplements during the trial period
* Able to understand research procedures and adhere to them throughout the entire study period
* Completed the run-in test

Exclusion Criteria:

* Diagnosis of dementia at a county-level or above hospital before the stroke or suspected to have pre-stroke dementia from the informant interview administered by a neurologist.
* Participation in or have participated in other clinical trial studies within the past year
* Allergies to foods involved in the experiment (nuts, berries, olive oil, or fish, etc.) or using drugs not compatible with foods involved.
* Medication to treat Alzheimer's or Parkinson's disease
* Diagnosis of cancer, severe liver and kidney disease, or current life expectancy less than 6 months
* Diagnosis of depression, bipolar disorder, or other mental illnesses
* Pregnancy or breastfeeding or with a pregnancy plan
* Diagnosis of inflammatory bowel disease or other malabsorption-related gastrointestinal diseases
* History of alcohol or drug abuse

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive function | 6 months
  Global cognitive function assessment is based on a battery of 18 cognitive tests. Individual test scores will be summarized by calculating the z-score for each test based on the mean and standard deviation of the sample distribution - averaging z-scores across tests will yield a composite score for global cognitive function. Cognitive function will be assessed at the baseline, 3, and 6 months to determine cognitive change.
Change in MIND diet score | 6 months
  Dietary behavior will be assessed using food frequency questionnaire (FFQ). A 15-point MIND diet score will be calculated to reflect the MIND diet adherence among both groups of participants.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score | 6 months
  MoCA will be administered at the baseline, 3, and 6 months to determine cognitive change.
Change in Mini-Mental State Examination (MMSE) score | 6 months
  MMSE will be administered at the baseline, 3, and 6 months to determine cognitive change.
Change in brain MRI markers | 6 months
  Changes in brain MRI-derived normalized measures of total brain volume (cubic centimetres) and hippocampal volume (cubic centimetres) and white/grey matter, segmented grey matter regions, white matter lesions, the thickness of segmented cortical regions, microbleeds, perivascular spaces, brain atrophy, micro-infarcts, and white matter hyperintensities. Change of functional connectivity measured using correlation coefficient of functional magnetic resonance imaging (fMRI) signal between brain regions. We will construct an overall brain health score as the outcome. Brain MRI will be assessed at the baseline and 6 months.
Change in memory function | 6 months
  Change in memory function will be assessed at the baseline, 3, and 6 months using the memory domain tests from the neuropsychological test battery.
Change in language function | 6 months
  Change in language function will be assessed at the baseline, 3, and 6 months using the language domain tests from the neuropsychological test battery.
Change in executive function | 6 months
  Change in executive function will be assessed at the baseline, 3, and 6 months using the executive function domain tests from the neuropsychological test battery.
Change in visuospatial function | 6 months
  Change in visuospatial function will be assessed at the baseline, 3, and 6 months using the visuospatial function domain tests from the neuropsychological test battery.

OTHER OUTCOMES:
Change in the ability of daily life measured using the Activities of Daily Living Scale (ADL) | 6 months
  To evaluate the effect on the ability of daily life of the MIND diet intervention. Evaluations will be conducted in 0, 3, and 6 months respectively.
Change in the ability of daily life measured using the Instrumental Activities of Daily Living Scale (IADL) | 6 months
  To evaluate the effect on the ability of daily life of the MIND diet intervention. Evaluations will be conducted in 0, 3, and 6 months respectively.
Change in depressive status measured using the Patient Health Questionnaire (PHQ-9) | 6 months
  To evaluate the effect on the depressive status of the MIND diet intervention. Evaluations will be conducted in 0, 3, and 6 months respectively.
Change in anxiety status measured using the General Anxiety Disorder-7 (GAD-7) | 6 months
  To evaluate the effect on the anxiety status of the MIND diet intervention. Evaluations will be conducted in 0, 3, and 6 months respectively.
Changes in plasma metabolic profiles measured using metabolome analysis | 6 months
  To evaluate the effect on plasma metabolites of the MIND diet intervention. We will assay the metabolome using liquid chromatography-mass spectrometry (LC-MS) and construct an overall metabolic score of the diet as the outcome. Evaluations will be conducted in 0 and 6 months respectively.
Changes in plasma inflammatory biomarker panel | 6 months
  To evaluate the effect on systematic inflammation of the MIND diet intervention. We will assay IFN-γ, interleukin (IL)-10, IL-12p70, IL-13, IL-1β, IL-2, IL4, IL6, IL-8, tumor necrosis factor (TNF)-α, and C reactive protein (CRP) and construct an overall plasma inflammatory biomarker score as the outcome. Evaluations will be conducted in 0 and 6 months respectively.
Changes in the intestinal microbiome | 6 months
  To evaluate the effect on intestinal microbiome biodiversity and abundance in specific species in faecal samples of the MIND diet intervention. We will assay microbiome using 16S ribosomal RNA (rRNA) sequencing and construct an overall intestinal microbiome score as the outcome. Evaluations will be conducted in 0 and 6 months respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Changzheng Yuan, ScD, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine; Lusha Tong, MD, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine; Xin Xu, PhD, Principal Investigator — Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Interested collaborators may put in a request.